CLINICAL TRIAL: NCT03235648
Title: Evaluation of Surgical Excision of Cardiophrenic Lymph Nodes in Patients With Advanced Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Basel Refky, MD, Doctor, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R/17.05.162
Record Dates: First submitted 2017-07-02; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cardiophrenic nodes excision in ovarian cancer (Experimental): We are going to evaluate the comorbidites and impact of cardiophrenic lymph nodes excision in cases of advanced ovarian cancer with positive cardiophrenic lymph nodes
  Interventions: Procedure: cardiophrenic lymph nodes resection

INTERVENTIONS:
Procedure: cardiophrenic lymph nodes resection — surgical resection

SUMMARY:
Evaluation of surgical excision of cardiophrenic lymph nodes in patients with advanced ovarian cancer

DETAILED DESCRIPTION:
The role of cardiophrenic lymph node assessment and excision in advanced ovarian cancer is still debatable , correlation of radiological finding with pathological findings after reaction of radiological positive lymph nodes and its impact in diseases free survival and over all survival

ELIGIBILITY:
Inclusion criteria

* Ovarian cancer patient (FIGO stage III-IV)
* Preoperative CT showing CPLN with short axis diameter > 5mm.
* Anathestically fit patient (ASA score I or II).
* Accepted pulmonary function test.
* Patient who received neoadjuvant chemotherapy or recurrent cases may be enrolled
* Written informed consent.
* Achievement of optimal cytoreduction intra-abdominal( No residual disease more than 1 cm )

Exclusion Criteria:

* Anathestically unfit patient
* Unresectable disease
* Patient refusal
* No detected CPLN by preoperative radiology

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
number of CPN retrieved/pathological nodes | up to 3 years
  correlation of radiological active lymph nodes with pathological findings

SECONDARY OUTCOMES:
Progression free survival | up to 2 years following the end of study
  2 years progression without disease recurrence

OTHER OUTCOMES:
Overall survival | up to 2 years following the end of study
  2 years survivals of the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology center, Mansoura University, Cairo, Dakhlia, Egypt

IPD SHARING:
Plan to Share IPD: No